CLINICAL TRIAL: NCT01386710
Title: Phase I/II Trial Of Repeated Super-selective Intraarterial Cerebral Infusion Of Bevacizumab Plus Carboplatin For Treatment Of Relapsed/Refractory Glioblastoma Multiforme And Anaplastic Astrocytoma
Brief Title: Repeated Super-selective Intraarterial Cerebral Infusion Of Bevacizumab Plus Carboplatin For Treatment Of Relapsed/Refractory GBM And Anaplastic Astrocytoma
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI left previous institution study will reopen at new institution.
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, John Boockvar, MD Zucker SOM @Hofstra/Northwell, MD, Feinstein Institute for Medical Research
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1012011410
Record Dates: First submitted 2011-06-13; First posted 2011-07-01 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma
Keywords: GBM; AA; AO; Brain; Tumors; Malignant; Glioblastoma; Multiforme; Anaplastic; Astrocytoma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Neoplasms | interventions — Bevacizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Arm 2 (Experimental): Drug: Bevacizumab and Carboplatin
  Interventions: Drug: Bevacizumab and Carboplatin
- Arm 1 (Experimental): Drug: Bevacizumab and Carboplatin
  Interventions: Drug: Bevacizumab and Carboplatin

INTERVENTIONS:
Drug: Bevacizumab and Carboplatin — Day 0: Intraarterial Bevacizumab single dose (15mg/kg) plus Intraarterial Carboplatin (150mg/m2) after Mannitol to open the blood brain barrier
  Day 28: Intravenous Bevacizumab (10mg/kg) plus Carboplatin (AUG5) every two weeks thereafter until disease progression on MRI scan.
  If progression occurs, repeat intraarterial Bevacizumab single dose (15mg/kg) plus intraarterial Carboplatin (150mg/m2) to area of progression and wait 28 days and then restart Intravenous Bevacizumab (10mg/kg) plus Carboplatin (AUG5) every two weeks thereafter until progression on MRI scan.
  Repeat Cycle
  Arms: Arm 1
Drug: Bevacizumab and Carboplatin — Day 0: Intraarterial Bevacizumab single dose (15mg/kg) plus Intraarterial Carboplatin (150mg/m2) after Mannitol to open the blood brain barrier
  Day 28: No biweekly IV Bevacizumab plus Carboplatin treatment
  If MRI shows progression then repeat intraarterial Bevacizumab single dose (15mg/kg) plus intraarterial Carboplatin (150mg/m2) to area of progression Repeat Cycle
  Arms: Arm 2

SUMMARY:
The high-grade malignant brain tumors, glioblastoma multiforme (GBM) and anaplastic astrocytoma (AA), comprise the majority of all primary brain tumors in adults. This group of tumors also exhibits the most aggressive behavior, resulting in median overall survival durations of only 9-12 months for GBM, and 3-4 years for AA. Initial therapy consists of either surgical resection, external beam radiation or both. All patients experience a recurrence after first-line therapy, so improvements in both first-line and salvage therapy are critical to enhancing quality-of-life and prolonging survival. It is unknown if currently used intravenous (IV) therapies even cross the blood brain barrier (BBB). The investigators have shown in a previous phase I trial that a single Superselective Intraarterial Cerebral Infusion (SIACI) of Bevacizumab (up to 15mg/kg) is safe and effective in the treatment of recurrent GBM. Therefore, this phase I/II clinical research trial is an extension of that trial in that the investigators seek to test the hypothesis that repeated dosing of intra-arterial Bevacizumab is safe and effective in the treatment of recurrent malignant glioma. Additionally the investigators will analyze if a combination with IA Carboplatin will further improve the treatment response. By achieving the aims of this study the investigators will also determine if IV therapy with Bevacizumab with IV Carboplatin should be combined with repeated selected intra-arterial Bevacizumab plus Carboplatin to improve progression free and overall survival. The investigators expect that this project will provide important information regarding the utility of repeated SIACI Bevacizumab therapy for malignant glioma, and may alter the way these drugs are delivered to the investigators patients in the near future.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Documented histologic diagnosis of relapsed or refractory glioblastoma multiforme (GBM), anaplastic astrocytoma (AA) or anaplastic mixed oligoastrocytoma (AOA).
* Circumscribed tumor recurrence with less than 3.5 cm greatest diameter
* Patients with histologically confirmed low-grade brain tumor relapse with an enhancing tumor on MRI will be evaluated for toxicity only.
* Patients must have at least one confirmed and evaluable tumor site.
* Patients must have a Karnofsky performance status 70% (or the equivalent ECOG level of 0-2)
* Patients must agree to use a medically effective method of contraception during and for a period of three months after the treatment period.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Patients with significant intercurrent medical or psychiatric conditions that would place them at increased risk or affect their ability to receive or comply with treatment or post-treatment clinical monitoring.
* Low GFR or history of hepatorenal syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2011-09; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Composite overall response rate | 6 months
  The composite overall response rate (CORR) will be examined. The overall response proportion along with a 95% confidence interval will be estimated via binomial proportions.
Six-month progression-free survival (PFS) and overall survival (OS) | 2 years
  PFS will be measured from the date of the first dose of SIACI Bevacizumab plus Carboplatin to the date of progression. OS will be measured from the date of the first dose of SIACI Bevacizumab plus Carboplatin to the date of death.

SECONDARY OUTCOMES:
The safety of repeated SIACI of Mannitol, Bevacizumab plus Carboplatin at 15mg/kg and 150mg/m2 respectively. | 1 month
  The descriptive frequency of subjects experiencing toxicities will also be tabulated. Toxicities will be assessed and graded according to the NCI Common Toxicity Criteria, version 3.0.

CONTACTS AND LOCATIONS:
Overall Officials: John Boockvar, MD, Principal Investigator — Lenox Hill Hospital
Locations (1):
- Lenox Hill Brain Tumor Center, New York, New York, United States

REFERENCES:
- See also: Drug Information available for: Bevacizumab — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0216974753&QV1=BEVACIZUMAB
- See also: Drug information for: Carboplatin — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0041575944&QV1=CARBOPLATIN